CLINICAL TRIAL: NCT05611463
Title: Camrelizumab Plus Docetaxel and Cisplatin as First-line Therapy in Recurrent or Metastatic Oral Squamous Cell Carcinoma Patients(CHANCE): an Open-label, Single-arm, Phase II Trial
Brief Title: Camrelizumab Plus Docetaxel and Cisplatin in Recurrent or Metastatic Oral Squamous Cell Carcinoma Patients
Acronym: CHANCE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SH9H-2019-T354-2
Record Dates: First submitted 2021-06-14; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-09

CONDITIONS: Oral Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — camrelizumab; Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab Plus Docetaxel and Cisplatin (Experimental): Participants receive Camrelizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle for up to 24 months;plus cisplatin 75 mg/m^2 IV or carboplatin at a target area under the curve of 5 (AUC 5) IV, per Investigator's choice, on Day 1 of each 3-week cycle (6 cycle maximum); plus docetaxel 75 mg/m^2 IV on Day 1 of each 3-week cycle (6 cycle maximum).
  Interventions: Drug: Camrelizumab Plus Docetaxel and Cisplatin

INTERVENTIONS:
Drug: Camrelizumab Plus Docetaxel and Cisplatin — Camrelizumab (200 mg) was administered once on day 1 every 3 weeks until disease progression, intolerable toxicity, physician or participant decision or 35 cycles, whichever occurred first. Chemotherapy was received docetaxel (75 mg/m2) and cisplatin (75 mg/m²) on day 2 every 3 weeks for six cycles.
  Other Names: SHR-1210+DTX+Platinol

SUMMARY:
the purpose of this study is to assess the efficacy and safety of camrelizumab plus Docetaxel and Cisplatin as First-line Therapy in Recurrent or Metastatic Oral Squamous Cell Carcinoma Patients

DETAILED DESCRIPTION:
Head and neck cancer is the sixth most common cancer in the world, with more than 550,000 cases and 300,000 deaths worldwide each year. About 75,000 Chinese suffer from head and neck cancer each year, and currently, there are a total of 176,000 patients with head and neck cancer in China. More than 95% of head and neck cancers are squamous cell carcinomas, and head and neck squamous cell carcinoma (SCCHN) disrupts and affects the patient's appearance and basic physiological functions, sensory functions, and language functions, thus affecting the patient's quality of life. Most head and neck squamous cell carcinomas are incurable, and they will develop local recurrence and metastasis.

More than 60% of patients with head and neck squamous cell carcinoma have stage III or IV disease characterized by large size tumors with marked local invasion, evidence of metastasis to regional lymph nodes, or both. Locally advanced head and neck cancer has a high risk of local recurrence and distant metastasis and a poor prognosis. Over the past 20 years, multimodal treatment approaches have steadily improved cure rates while striving to maintain patient function and quality of life.

This clinical study involved Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection (Camrelizumab), a Class 1 new therapeutic biological product developed by Jiangsu Hengrui Medicine Co., Ltd., which was approved by NMPA in May 2019 for the treatment of relapsed or refractory classical Hodgkin's lymphoma, by NMPA in March 2020 for the treatment of patients with advanced hepatocellular carcinoma who have received sorafenib and/or oxaliplatin-based systemic chemotherapy, and in June 2020 for the second-line treatment of esophageal squamous cell carcinoma and first-line treatment of non-squamous non-small cell lung cancer.

Preclinical study data showed that camrelizumab had comparable in vivo efficacy and safety compared with similar drugs abroad. Since 2015, Hengrui has simultaneously carried out a number of phase I/II clinical trials in Australia and China to preliminarily verify the safety, tolerability and efficacy of camreibizumab in the treatment of advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed post-surgical recurrent/metastatic or locally advanced inoperable oral squamous carcinoma with measurable lesions (spiral CT scan ≥ 10 mm, meeting RECIST 1.1 criteria).
* No prior treatment with any systemic antineoplastic agent, prior adjuvant or neoadjuvant therapy (other than PD-1/PDL-1 monoclonal antibody) is allowed, provided that it was completed at least 4 weeks prior to the first dose of study drug and all associated toxic events have returned to normal or to grade I or below as defined by CTCAE 4.03 classification.
* An ECOG score of 0 or 1.
* Expected survival of ≥ 12 weeks.
* Normal function of major organs within 2 weeks prior to treatment, i.e. meeting the following criteria.

Bone marrow function: hemoglobin ≥ 100gg/L, white blood cell count ≥ 4.0*10^9/L or neutrophil count ≥ 2.0*10^9/L and platelet count ≥ 100*10^9/L without transfusion or with colony-stimulating factor support therapy.

Liver: serum total bilirubin level ≤ 1.5 times the upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 1.5 times the upper limit of normal.

Renal: blood creatinine level less than 1.5 times the upper limit of normal or creatinine clearance ≥ 60 ml/min and urea nitrogen ≤ 200 mg/L. Urine protein <+, if urine protein + then total 24 hour protein must be <500mg.

Blood glucose: within normal range and/or with diabetic patients on treatment but with stable blood glucose control.

Pulmonary function: baseline FEV1 of at least 2L, if baseline FEV1 < 2L, FEV1 >800ml is expected after surgery as assessed by a surgical specialist.

Cardiac function: no myocardial infarction within 1 year; no unstable angina; no symptomatic severe arrhythmia; no cardiac insufficiency.

* Women of childbearing potential must have a negative serum pregnancy test result within 7 days prior to the first dose of the test drug; men of childbearing potential or women of childbearing potential must use a highly effective contraceptive method (e.g., oral contraceptive pill, intrauterine device, abstinence from sexual intercourse, or barrier contraceptive method combined with spermicide) throughout the trial and continue to use contraception for 12 months after the end of treatment.

Exclusion Criteria:

* Patients with prior anti-PD-1, anti-PD-L1, anti-PD-L2 therapy. Patients who are currently receiving antineoplastic therapy.
* Patients who have participated or are participating in a clinical trial of another drug/therapy within 4 weeks prior to the first dose of the study drug.
* Patients with any active autoimmune disease or history of autoimmune disease (e.g., the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enterocolitis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism; patients with vitiligo; asthma that has completely resolved in childhood and does not require any intervention in adulthood may be included; patients who require medical intervention with bronchodilators (asthma, on the other hand, cannot be included).
* Patients who are on immunosuppressive, or systemic hormone therapy for immunosuppressive purposes (doses >10 mg/day prednisone or other equipotent hormone) and are continuing to use them within 2 weeks prior to enrollment.
* Patients who have received hematopoietic stimulating factors, such as granulocyte colony-stimulating factor (G-CSF), erythropoietin, etc., within 1 week prior to the first administration of the study drug.
* Positive test results for HIV antibodies or syphilis spirochete antibodies. Patients with active hepatitis B or C:
* If HBsAg or HBcAb is positive, add HBV DNA test (the result is higher than the upper limit of the normal range).
* Additional HCV RNA testing if positive for HCV antibodies (results above the upper limit of the normal range).
* Persons with known hypersensitivity to recombinant humanized PD-1 monoclonal antibody drugs and their components.
* Massive pleural or ascites fluid with clinical symptoms and requiring symptomatic management.
* Active lung disease (interstitial pneumonia, pneumonia, obstructive lung disease, asthma) or a history of active tuberculosis.
* Have any clinical problems beyond their control, including but not limited to: Persistent or active (severe) infection;
* Poorly controlled diabetes;
* Cardiac disease (Class III/IV congestive heart failure or heart block as defined by the New York Heart Association);
* Have or suspect autoimmune disease, or a history of autoimmune disease or syndrome requiring steroid/immunosuppressive systemic therapy, such as: hypopituitaritis, colitis, hepatitis, nephritis, hyperthyroidism, hypothyroidism, etc;
* Deep vein thrombosis or pulmonary embolism; myocardial infarction; severe or unstable arrhythmia or angina; percutaneous coronary intervention, acute coronary syndrome, coronary artery bypass grafting; cerebrovascular accident, transient ischemic attack, cerebral embolism within 6 months prior to first dose.
* Abnormal coagulation (INR > 2.0, PT > 16s), with bleeding tendency or on thrombolytic or anticoagulant therapy, allowing prophylactic use of low-dose aspirin, low-molecular heparin.
* Those who had clinically significant bleeding symptoms or clear bleeding tendency within 3 months prior to randomization, such as daily cough/hemoptysis of 2.5 ml or more, gastrointestinal bleeding, esophagogastric fundic varices at risk of bleeding, bleeding gastric ulcers or suffering from vasculitis, etc., may be reviewed if the fecal occult blood is positive at baseline, and if it is still positive after review, gastroscopy is required, and if gastroscopy indicates severe esophagogastric fundic varices cannot be enrolled (except for those who underwent gastroscopy 3 months or less before enrollment to exclude such conditions).
* Known presence of hereditary or acquired bleeding and thrombotic tendencies (e.g., hemophiliacs, coagulation disorders, thrombocytopenia, etc.)
* Have received a stem cell transplant or organ transplant.
* Those with a history of psychotropic substance abuse and unable to abstain or a history of mental disorders.
* Other serious, acute or chronic medical conditions or laboratory test abnormalities that, in the judgment of the investigator, may increase the risk associated with participation in the study, or may interfere with the interpretation of study results.
* The patient had a history of other malignancies within five years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-06-02 (Actual); Primary Completion 2022-12-02 (Estimated); Study Completion 2023-06-02 (Estimated)

PRIMARY OUTCOMES:
Participants Experiencing an Adverse Event (AE) | 24 months
  An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The number of participants that experienced at least one AE was reported for treatment arm

SECONDARY OUTCOMES:
Objective remission rate (ORR) | 24 months
  radiographically confirmed complete or partial response
overall survival | 24 months
  the time from enrolled to death from any cause
progression -free survival | the time from enrolled to radiographically confirmed disease progression or death from any cause (whichever occurred first)
  the time from enrolled to radiographically confirmed disease progression or death from any cause (whichever occurred first)
Duration of remission (DOR) | 24 months
  the time from first documented complete or partial response to radiographically confirmed disease progression or death from any cause, whichever occurred first

CONTACTS AND LOCATIONS:
Overall Officials: Yue He, M.D., Principal Investigator — the Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Ninth People's Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No